CLINICAL TRIAL: NCT01986192
Title: An Efficacy and Safety Study of Ribaroxaban for the Prevention of Deep Vein Thrombosis Recurrence in Patients With Acute Iliofemoral Venous Thrombosis Initially Treated With Thrombolysis
Brief Title: Prevention of Recurrence After Thrombolysis in Acute Iliofemoral Venous Thrombosis (PRAIS) Study
Acronym: PRAIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Daegu Catholic University Medical Center (Other); Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Seung-Kee Min, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRAIS-1.1-12-12
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Ileofemoral Deep Vein Thrombosis
Keywords: anticoagulation; pharmacomechanical thrombolysis; aspiration thrombectomy
MeSH Terms: interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rivaroxaban (Experimental): Rivaroxaban 15mg bid for 3 weeks and 20mg qd for 6 months
  Interventions: Drug: rivaroxaban
- warfarin (Active Comparator): Enoxaparin 1mg/kg bid overlapping with warfarin (target PT INR 2.0-3.0) for 6 months
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: rivaroxaban
  Other Names: xarelto
  Arms: rivaroxaban
Drug: Warfarin
  Arms: warfarin

SUMMARY:
The EINSTEIN program showed that oral rivaroxaban is effective and safe treatment for prevention of recurrent venous thrombosis and pulmonary embolism in deep vein thrombosis patients and FDA approved the rivaroxaban for prevention and treatment of deep vein thrombosis (Nov 2 2012).

Recently, catheter-directed thrombolysis can significantly reduce post-thrombotic syndrome, and more and more centers introduce catheter-directed thrombolysis to treat proximal (i.e, iliofemoral) DVT. However, the EINSTEIN program excluded patients with deep vein thrombosis if they had been treated with a vena cava filter or a fibrinolytic agent for the current episode of thrombosis.

Although catheter-directed thrombolysis (CDT) or pharmacomechanical thrombolysis has now been accepted as a treatment of choice in iliofemoral DVT, thrombolysis has an inherent risk of bleeding. Therefore, patients who have completed CDT and have been stabilized at least 24 hours after thrombolysis will be included in this study.

Also, the investigators want to explore the efficacy and safety of rivaroxaban in patients with iliofemoral DVT after catheter-directed thrombolysis and/or a vena cava filter insertion and/or venous stent insertion and compare these outcomes with warfarin treatment alone.

This study will be a pilot study to establish the safety and efficacy parameters for further studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Onset of symptoms within the past 21 days
* Objectively verified (by CT venography) deep vein thrombosis localized in the iliofemoral segment
* Complete catheter-directed thrombolysis and/or a vena cava and/or venous stent insertion
* Informed consent

Exclusion Criteria:

* Incomplete catheter-directed thrombolysis
* If patients received more than a single dose of a warfarin before randomization
* contraindicating anticoagulant treatment
* another indication for a warfarin
* an estimated glomerular filtration rate by MDRD equation <30ml/min
* clinically significant liver disease (acute hepatitis, chronic active hepatitis, cirrhosis)
* Alanine aminotransferase > 3-time higher than upper limit of the normal range
* Bacterial endocarditis
* Active bleeding or high risk of bleeding
* Pregnancy or breast-feeding
* Concomitant use of strong cytochrome P-450 3A4 inhibitors or inducers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-02 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | six month
  to compare recurrence rate within 6 months after thrombolysis in iliofemoral deep vein thrombosis with warfarin prophylaxis

SECONDARY OUTCOMES:
vascular events | six months
  All-cause mortality, vascular events (acute coronary syndrome, ischemic stroke, transient ischemic attack or systemic embolism)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Kee Min, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea